CLINICAL TRIAL: NCT04752072
Title: RESTORE Trial: A Pilot RCT of Enhanced Skills Training in Affective and Interpersonal Regulation (ESTAIR) vs. Treatment as Usual (TAU) for Complex Posttraumatic Stress Disorder (CPTSD) in Military Personnel
Brief Title: RESTORE Trial: A Pilot RCT of Enhanced Skills Training in Affective and Interpersonal Regulation (ESTAIR) for Veterans With CPTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Combat Stress (Other)
Collaborators: Edinburgh Napier University (Other)
Responsible Party: Principal Investigator, Prof. Dominic Murphy, Head of research department, Combat Stress
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHSC2686062; FiMT19/0429EDU (Other Grant/Funding Number: Forces in Mind)
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Complex Post-Traumatic Stress Disorder
Keywords: CPTSD; ESTAIR; modular therapy
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to the intervention arm (ESTAIR) or the control arm (TAU)
Who Masked: Outcomes Assessor
Masking Description: It was initially intended for the research assistant collecting post-intervention and follow-up outcome measures to be masked to arm allocation. However, it is noted that such masking is not feasible. This is not deemed a risk to the study as outcome measures are self-report measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESTAIR (Experimental): ESTAIR (Cloitre et al., 2019) will consist of up to 25 sessions, organized in 4 modules of 6 sessions targeting symptoms of PTSD and disturbances in self-organisation (AD: affective dysregulation; NSC: negative self-concept; and DR: disturbances in relationships).
  Interventions: Behavioral: Enhanced Skills Training in Affective and Interpersonal Regulation
- Treatment as usual (TAU) (Active Comparator): At present, there are no recommended treatments for CPTSD. TAU will consist of a treatment package that could include elements of psychoeducation, symptom-management and trauma-focused cognitive behaviour therapy, resembling established protocols for treating PTSD.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Enhanced Skills Training in Affective and Interpersonal Regulation — The first (formulation) session enables linking present difficulties and traumatic events, identifying current issues/concerns, and collaboratively agreeing on the order of modules based on symptom severity and client readiness.
  The PTSD module provides narrative exposure to the traumatic memories and targets re-experiencing, avoidance and hyperarousal symptoms. The AD module focuses on identifying and labelling feelings, emotion management, distress tolerance, acceptance of feelings and experiencing positive emotions. The NSC module focuses on staying in the present moment and combating dissociation; self-compassion and mindfulness skills; challenging thinking patterns and developing a balanced view of self. The DR module focuses on exploring and revising maladaptive schemas; effective assertiveness; awareness of social context; and flexibility in interpersonal expectations and behaviours displayed in social interactions.
  Arms: ESTAIR
Behavioral: Treatment as usual — The first session will involve a mental health assessment by either a psychiatrist or psychologist. A treatment package will be developed based on the information collected during the assessment. Details of the interventions delivered to each participant receiving TAU, which will include elements of psychoeducation, symptom-management and trauma-focused cognitive behaviour therapy, will be recorded.
  Arms: Treatment as usual (TAU)

SUMMARY:
Complex Post traumatic Stress Disorder (CPTSD) is now recognized as a separate trauma-based psychological condition to PTSD. CPTSD is a broader diagnosis that includes the core PTSD symptoms (re-experiencing in the here and now, avoidance, and sense of current threat) plus an additional set of symptoms that are collectively referred to as 'disturbances in self-organisation' (DSO). DSO symptoms capture pervasive psychological disturbances that are associated with traumatic exposures and that are distributed across three clusters: difficulties in affect regulation (AR), negative self-concept (NSC), and disturbances in relationships (DR).

There are no effective interventions for CPTSD. It is therefore of paramount important to identify effective interventions to treat veterans with CPTSD. The present study will be one of the first to investigate the effectiveness of a novel, modular intervention for CPTSD. Enhanced Skills Training in Affective and Interpersonal Regulation (ESTAIR) is a person-centered intervention that involves targeting the symptoms of CPTSD clusters sequentially using concrete modules (i.e., specific number of sessions targeting specific clusters of symptoms).

The overall aim of this study is to establish the feasibility, acceptability and preliminary effects of ESTAIR in treating CPTSD. To achieve these aims, the investigators will conduct a pilot randomised controlled trial (RCT), with a sample of 60 military veterans meeting the diagnostic criteria for CPTSD, and with two treatment arms: ESTAIR vs. a treatment-as-usual (TAU) condition.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) in the caseload of Combat Stress
* Armed forces veteran (United Kingdom)
* Help-seeking for trauma-related psychological distress
* Meeting diagnostic criteria for CPTSD, as measured by the ITQ (Cloitre et al., 2018)
* Proficiency in English language
* Signed informed consent provided

Exclusion Criteria:

* Severe psychotic disorder (defined by previous clinical diagnosis)
* Current alcohol or drug use disorder
* Serious cognitive impairment
* Planned concurrent additional treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Retention rate at the end of treatment | Post-treatment (week 25)
  Percentage of clients completing intervention and completing outcome measures at the end of treatment.
Retention rate at 3-months follow up | 3-months follow-up (week 37)
  Percentage of clients completing intervention and completing outcome measures at 3-months follow up.
Change in symptoms of CPTSD on the International Trauma Questionnaire (ITQ) from baseline to end of treatment to 3-months follow up | Baseline, end of treatment (week 25) and 3-months follow up (week 37)
  The ITQ (Cloitre et al., 2018) is a validated questionnaire assessing PTSD and complex-PTSD (CPTSD). Six items represent the three clusters of PTSD (re-experiencing, avoidance and sense of threat), while another six items represent the three clusters reflecting disturbances in self-organisation (DSO) (AD: affective dysregulation; NSC: negative self-concept; and DR: disturbances in relationships. The remaining items assess functional impairment relating to symptoms of PTSD (3 items) and DSO (3 items). Items are scored using 5-point Likert scales ranging from 0 (not at all) to 4 (extremely), indicating how much a symptom has affected them in the past month.
  A diagnosis of CPTSD required a diagnosis of PTSD (at least one symptom of each of its three clusters as well as functional impairment) in addition to endorsement of at least one symptom of each of the three DSO clusters plus functional impairment.

SECONDARY OUTCOMES:
Change in symptoms of depression on the 9-item Patient Health Questionnaire (PHQ-9) from baseline to end of treatment to 3-months follow up | Baseline, end of treatment (week 25) and 3-months follow up (week 37)
  The PHQ-9 (Korienke et al., 2001) is a 9-item questionnaire of depression. Items are scored using 4-point Likert scales ranging from 0 (not at all) to 3 (nearly every day), indicating how much they have been bothered by a symptom over the past two weeks. Total scores range from 0 to 27, with higher scores indicating greater levels of depression. Cut-off scores of 15 are used to identify participants likely meeting criteria for depressive disorder.
Change in symptoms of generalised anxiety on the 7-item Generalised Anxiety Disorder Questionnaire (GAD-7) from baseline to end of treatment to 3-months follow up | Baseline, end of treatment (week 25) and 3-months follow up (week 37)
  The GAD-7 (Spitzer et al., 2006) is a 7-item questionnaire of generalised anxiety. Items are scored using 4-point Likert scales ranging from 0 (not at all) to 3 (nearly every day), indicating how much they have been bothered by a symptom over the past two weeks.
  Total scores range from 0 to 21, with higher scores indicating greater levels of anxiety. Cut-off scores of 10 are used to identify participants likely meeting criteria for generalised anxiety disorder.
Change in alcohol use on the 3-item (AUDIT-C) from baseline to end of treatment to 3-months follow up | Baseline, end of treatment (week 25) and 3-months follow up (week 37)
  The AUDIT-C (Saunders et al., 1993) consists of the first three items of the Alcohol Use Disorders Identification Test. Items are scored using a 4-point Likert scale. Total scores range from 0 to 12. Based on a nationally representative sample of adults from the United States, scores ≥ 4 effectively capture a diagnosis of Alcohol Use Disorder (AUD).
Change in medically unexplained symptoms on the 15-item Patient Health Questionnaire-15 (PHQ-15) from baseline to end of treatment treatment to 3-months follow up | Baseline, end of treatment (week 25) and 3-months follow up (week 37)
  The PHQ-15 (Korienke et al., 2002) is a 15-item questionnaire of somatisation disorder symptoms. Items are scored using 4-point Likert scales ranging from 0 ("not bothered at all") to 3 ("bothered a little" or "nearly every day"), indicating how much they have been bothered by a symptom over the past two weeks. Total scores range from 0 to 30, with scores of of ≥5, ≥10, ≥15 representing mild, moderate and severe levels of somatization.
Outcome on the single item Friends and Family Test (FFT) at end of treatment. | End of treatment (week 25)
  The FFT is a single item assessing the acceptability of an intervention (i.e., ' How likely is it that you would recommend our service to your GP, family and friends if they needed similar care?'). The item is scores on a 5-point Likert scale ranging from 1 ("extremely unlikely") to 5 ("extremely likely". The FFT is standardly administered as an end-of-treatment measure at Combat Stress

OTHER OUTCOMES:
Experience of potentially traumatic life events on the Life Events Checklist (LEC) | Baseline
  The LEC (Gray et al., 2004) is a 17-item questionnaire assessing potentially traumatic events in the respondent's lifetime. The LEC assesses exposure to 16 events plus one item assessing any other extraordinary stressful event. Respondents report whether they 1) directly experienced, 2) witnessed, 3) learned about, 4) are not sure, or 5) does not apply to them.
Rates of adverse events at end of treatment and 3-months follow up | End of treatment (week 25) and 3-months follow up (week 37)
  Using a previously applied approach (adapted from Klingberg et al., 2012), we will define serious adverse events as (i) death by suicide; (ii) suicide attempt; (iii) suicidal crisis without attempt; (iv) severe symptom exacerbation (increase of 2 standard deviations or more on the patient or researcher-rated ITQ. Non-severe adverse events will be defined as a score of ≥3 (agree 'quite a lot' or 'a lot') on any relevant item (e.g., subjectively worsening mental state, heightened stigma, increased medication use, increased conflict) on the patient-rated Adverse Events Questionnaire (adapted from Hutton et al., 2015).
  Participants who withdraw from the study will also be asked to complete the Adverse Events Questionnaire (adapted from Hutton et al., 2015) to determine whether withdrawal is due to adverse events.
Change in symptoms of CPTSD on the International Trauma Questionnaire (ITQ) following each module in ESTAIR arm only | Week 7, Week 13, Week 19, Week 25
  The ITQ (Cloitre et al., 2018) is described above as the primary outcome measure. Six items represent the three clusters of PTSD. Another six items represent the three clusters reflecting disturbances in self-organisation (DSO). The remaining items assess functional impairment relating to symptoms of PTSD (3 items) and DSO (3 items). Items are scored using 5-point Likert scales ranging from 0 (not at all) to 4 (extremely), indicating how much a symptom has affected them in the past month.
  The ITQ will be completed following each module in the ESTAIR arm to gain insight into the progression of CPTSD symptoms during treatment and to support discontinuation of treatment should any adverse symptom exacerbation occur.
Change in symptoms of the moral injury on the 14-item Moral Injury Outcome Scale (MIOS) from baseline to 3-months follow-up | Baseline and 3-months follow up (week 37)
  The MIOS (Litz et al., 2020) is a 14-item questionnaire of moral injury. Items are scored using 5-point Likert scales ranging from 0 (strongly disagree) to 3 (strongly agree), indicating how much they would agree with each statement in the past month. Total scores range from 0 to 60, with higher scores indicating greater severity of moral injury.
  *Due to further validation work, the MIOS has been amended from a 15-item measure to a 14-item measure of moral injury.
Qualitative data regarding acceptability of the ESTAIR intervention (ESTAIR arm only) | End of treatment (Week 25)
  Participants completing the ESTAIR intervention will have a one-off interview to collect information regarding their experiences of treatment in general, the protocol, and overall participation.
  Client will provide their subjective experience of the intervention, including positive and negative aspects of the treatment, the impact on their wellbeing, and be asked to offer suggestions for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Murphy, Prof., Principal Investigator — Combat Stress; Thanos Karatzias, Prof., Principal Investigator — Edinburgh Napier University
Locations (1):
- Combat Stress, Leatherhead, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data collected in this study will be stored for 10 years and will not be made available to other researchers (because of the small sample sizes involved).
  Summary data will be provided in publications, but the individual data will not be available given the risks this raises with identification of participants.
  The data will not be shared except for the purposes of audit by Edinburgh Napier University or Combat Stress approved staff.

REFERENCES:
- [Background] Cloitre, M., Karatzias, T., Mc Glanaghy, E. (2019). Enhanced STAIR Narrative Therapy for CPTSD. Treatment Manual. Unpublished Manuscript.
- [Background] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Gray MJ, Litz BT, Hsu JL, Lombardo TW. Psychometric properties of the life events checklist. Assessment. 2004 Dec;11(4):330-41. doi: 10.1177/1073191104269954. PMID 15486169
- [Background] Hutton P, Byrne R, Pyle M, Morrison AP. Adverse Effects of Psychological Therapy Questionnaire. Unpublished; 2015.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT04752072/Prot_SAP_003.pdf